CLINICAL TRIAL: NCT03955302
Title: Ultrasound Assessment of Muscle Architecture Before and After the Implementation of a Physical Exercise Regime in the Water in a Frail Elderly Population
Brief Title: Ultrasound Assessment of a Physical Exercise in The Water in a Frail Population
Acronym: SWIMFRAIL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1557856842051
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2019-05

CONDITIONS: Frailty Syndrome
Keywords: Frailty; Muscle Architecture; Ultrasound; Exercise Regimen; Aqua-Aerobics
MeSH Terms: conditions — Frailty | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Patients in this group will perform the water exercise protocol, 3 times a week, for 12 weeks.
  Interventions: Behavioral: Exercise
- Control (No Intervention): Patients in this group will not perform any type of exercise during the 12 weeks of the treatment.

INTERVENTIONS:
Behavioral: Exercise — There will be an intervention for 12 weeks. For exercises in the water, there will be an expert physiotherapist in the field of hydrotherapy that will guide the exercises in controlled sessions of approximately 45 minutes. Exercises of joint mobility, balance, strength and coordination with / without aquatic material will be included. At all times, qualified health personnel will monitor any symptom or sign that advises the removal of the subject of the study.
  Arms: Exercise

SUMMARY:
It is an experimental, longitudinal prospective, controlled trial. The project will be developed in the General University Hospital of Valencia (CHGUV), and the University of Valencia.

Patients will be recruited from a previous cohort. The patients of this cohort will be contacted and proposed to participate. Those patients who accept, will be divided into the following experimental groups:

* Group 1: Patients in this group will perform the water exercise protocol, 3 times a week, for 12 weeks.
* Group 2: Patients in this group will not perform any type of exercise during the 12 weeks of the treatment.

Variables related to muscular quality by ultrasound, frailty, physical function, independence in the activities of daily life, balance, cognitive function, quality of life and sleep, the social sphere will be evaluated, and the intensity of pain and fatigue, before and after12 weeks of intervention.

DETAILED DESCRIPTION:
OBJECTIVE To evaluate changes in muscle architecture by ultrasound, before and after an intervention with physical exercise directed in water in frail individuals; and determine the correlation of the image findings with the changes detected in their morbidity, functionality and quality of life.

SAMPLE

The sample will be composed of at least 40 frail men and women, according to Frail Phenotype criteria. Patients will be recruited from a previous cohort. For the assessment of frail, Linda Fried's criteria will be used: unintentional weight loss, feeling of general exhaustion, slow gait, low level of physical activity or muscular weakness. A point will be assigned to each positive criterion. A final score formed by the sum of the five criteria. According to this score, subjects will be classified as follows:

* Non-frail: 0 points
* Pre-frail: 1 or 2 points
* Frail: 3 or more points

STUDY DESIGN It is an experimental, prospective, controlled study. Patients will be recruited from a previous cohort performed at the General University Hospital of Valencia (CHGUV). This study was entitled "Muscular architecture study by ultrasound for the diagnosis of frail with correlation of clinical, physical and biochemical markers". The patients of this cohort will be contacted by telephone, where they will be proposed to participate in the present study. Patients that accept will be ask to undergo a muscle ultrasound. At that time those who meet the inclusion criteria and none of the exclusion criteria, will be presented with the option of participating in the targeted exercise intervention. The subjects will be divided into Group 1 (Exercise) or Group 2 (Control). Those who agree to participate will be given the informed consent, offering them the appropriate time to read it and resolve doubts about it.

All eligible subjects will be informed of the objectives of the study and will be asked to collaborate in it. Before the ultrasound examination, the patients will be explained that the procedure is experimental and what is the purpose of the study. Being a study with intervention, the need to maintain maximum adherence to the physical exercise regime during the 12 weeks, as well as the need to perform all assessments both before and after the intervention.

Variables related to the diagnosis of muscular quality by ultrasound, frailty condition, morbidity, physical function, independence in the activities of daily life, balance, cognitive function, quality of life and sleep, the social sphere will be evaluated, and the intensity of pain and fatigue, before and after the 12 weeks of intervention.

The muscular ultrasound will be performed in the Radiology Department of the Hospital. At the conclusion of the ultrasound, a muscle strength measurement will be performed with a dynamometer and patients will fill out a questionnaire of epidemiological data, medical history, comorbidities and, criteria of frailty. A second appointment will be scheduled to make a blood extraction for biochemical analysis. After concluding the intervention, patients will be called again to perform a follow-up ultrasound, questionnaires, physical function assessment and biochemical analysis.

INTERVENTION For the exercise in the water (aqua aerobics), there will be an expert physiotherapist in the field of hydrotherapy that will guide the exercises in controlled sessions of approximately 45 minutes. Exercises of joint mobility, balance, strength and coordination with / without aquatic material (tables, cork anklets, long corks, cork dumbbells, pull-boy, and inflatable collars, among others) will be included. At all times, qualified health personnel will monitor any symptom or sign that advises the removal of the subject of the study (maintained dizziness, hypertension or uncontrolled hypotension, chest pain, muscular or tendon injuries, etc).

MUSCULAR ULTRASOUND Studies of muscle architecture through ultrasound show a non-invasive method to detect isometric contraction of individual muscles. In addition to being non-invasive, accessible and economical, it allows the dynamic exploration of the muscle under study.

The ultrasound allows, on the one hand, assessment of the quantitative parameters at rest and contraction, measuring muscle thickness, anatomical and physiological area puncture angle and fascicular length. On the other hand, muscle intensity echo will be assessed as a qualitative parameter. The muscle architecture of the anterior compartment of the leg will be evaluated by ultrasound in B mode, obtaining transverse and longitudinal images with a linear transducer (6-15 MHz). The measurements of the muscle ultrasound will be made three times and the average of said measurements will be used in the data analysis. The images made during the scan will be stored in the hospital picture archiving and communication system (PACS).

DATA COLLECTION The first section of the questionnaire will include questions about general epidemiological data and details of the patient's medical history. The following parameters will be recorded: age, gender, marital status (single, married or widowed) and social situation (spouse, alone or with children). Among the anthropometric parameters, the height and the weighed of the participants will be measured to perform the calculations of the patient's body mass index. The presence or absence of hypertension, hyperlipidemia, diabetes mellitus, heart failure according to Framingham criteria, ischemic heart disease, presence of previous stroke, chronic obstructive disease, smoker (yes, no or ex-smoker) will be included in the patient's clinical history. Visual problems, hearing problems, Parkinson's disease, depression, previous cancer, kidney failure, arthritis, osteoporosis and number of recent fractures will also be assessed. In addition, an index of comorbidities will be carried out according to the Charlson index using an online calculator and number of falls in the previous 6 months. And finally, the number of visits to the primary care physician, emergencies and hospital admissions in the last 6 months.

ASSESSMENT OF PHYSICAL FUNCTION Various tests will be carried out to assess the physical function. Individuals will be asked the following requirements: comfortable clothing and footwear, light food (no fasting prior to the test), no intense exercise in the previous 2 hours, no present conditions that limit walking, and that may interfere with the interpretation of the test, such as injuries to the lower extremities or respect the schedules of the medication that the patient takes regularly. All tests will be conducted by a qualified physiotherapist. The test are 6-minute walk test, Borg Scale, Short Physical Performance Battery (SPPB), and "timed up and go" test. Likewise, different scales will be carried out to assess the independence, and activities of daily life, assessment of balance or risk of falls. For the assessment of cognitive function (Hospital Anxiety and Depression Scale (HADS), for the assessment of quality of life (Older People Quality of Life (OPQOL), and sleep (Pittsburgh Sleep Quality Index), for the assessment of the social sphere (Duke social support), and for the assessment of pain intensity (McGill Questionnaire) and fatigue (fatigue severity scale).

BIOCHEMICAL BIOMARKERS A blood extraction will be requested by the subjects general practitioners. A blood sample will be taken from the CHGUV clinical analysis department before and after the intervention. The biomarkers will be measured in a blood sample drawn between 8:00 a.m. and 10:30 a.m. after fasting for at least 8 hours and your usual procedure will be done with the protocols already established in the bio clinical analysis department.

STATISTICAL ANALYSIS The descriptive data are presented with the mean ± standard deviation (SD) with the distribution of the data verified by the Shapiro-Wilk and / or Kolmogorov-Smirnov normality test. To evaluate differences in physical characteristics and study variables, t-Student was used for parametric and Mann-Whitney variables for non-parametric variables. The evaluation of the different study variables according to the stages of fragility and control group will be determined by means of analysis of variance (ANOVA) for the parametric variables (followed by the Bonferroni post hoc test) and for the non-parametric Kruskal-Wallis test. To assess the sonographic changes after the intervention of the patients with directed exercise, the T-student test will be used for paired data. The correlations will be made with the Pearson coefficient for parametric data and the Spearman range for non-parametric data. The correlations were considered weak for the correlation coefficient of ± 0.01 to 0.35, moderate for ± 0.36 to 0.67 and strong for ± 0.68 to 1.00. To compare the reliability between sonographer and evaluators of functional tests; we perform the intraclass correlation coefficient (ICC) and the Bland-Altman agreement limits of 95%. The ICC values were classified as poor for values ≤0.20, just for 0.21-0.40, moderate for 0.41-0.60, good for 0.61-0.80 and very good for 0.81-1.00. To assess the accuracy of muscle ultrasound, the area under the receiver operating characteristic (ROC) curve or curves will be determined. The statistical significance will be defined a priori as P <0.05. All statistical analyses will be performed with Statistical Package for the Social Sciences (SPSS) version 24.0 for Windows.

ELIGIBILITY:
Inclusion Criteria:

* Age between 65 and 95 years, be physically inactive (<150 min physical activity a week), meet 1 or more criteria of frailty according to Linda Fried criteria, signature of informed consent.

Exclusion Criteria:

* Institutionalized patients, life expectancy of less than 6 months for any reason, hospital admission in the last 3 months for any reason; major surgery in the last 6 months before the start of the study, oncological patient with active treatment with chemotherapy or radiotherapy; neurological or musculoskeletal pathology that contraindicates physical activity in water; severe disability (score below 15 points on the Barthel scale); severe cardiovascular disease, psychotic disorder or severe cognitive impairment.

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Muscle Architecture Improvement | 14 weeks
  Muscle measurement with ultrasound before and after the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Consuelo M Borras Blasco, PhD, Study Director — University of Valencia
Locations (1):
- Hospital General Universitario de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abe T, Loenneke JP, Thiebaud RS, Fukunaga T. Age-related site-specific muscle wasting of upper and lower extremities and trunk in Japanese men and women. Age (Dordr). 2014 Apr;36(2):813-21. doi: 10.1007/s11357-013-9600-5. Epub 2013 Nov 17. PMID 24243442
- [Result] Arts IM, Pillen S, Overeem S, Schelhaas HJ, Zwarts MJ. Rise and fall of skeletal muscle size over the entire life span. J Am Geriatr Soc. 2007 Jul;55(7):1150-2. doi: 10.1111/j.1532-5415.2007.01228.x. No abstract available. PMID 17608902
- [Result] Arts IM, Pillen S, Schelhaas HJ, Overeem S, Zwarts MJ. Normal values for quantitative muscle ultrasonography in adults. Muscle Nerve. 2010 Jan;41(1):32-41. doi: 10.1002/mus.21458. PMID 19722256
- [Result] Bouillon K, Kivimaki M, Hamer M, Sabia S, Fransson EI, Singh-Manoux A, Gale CR, Batty GD. Measures of frailty in population-based studies: an overview. BMC Geriatr. 2013 Jun 21;13:64. doi: 10.1186/1471-2318-13-64. PMID 23786540
- [Result] Bowling A. The Psychometric Properties of the Older People's Quality of Life Questionnaire, Compared with the CASP-19 and the WHOQOL-OLD. Curr Gerontol Geriatr Res. 2009;2009:298950. doi: 10.1155/2009/298950. Epub 2010 Feb 1. PMID 20168974
- [Result] Bressel E, Wing JE, Miller AI, Dolny DG. High-intensity interval training on an aquatic treadmill in adults with osteoarthritis: effect on pain, balance, function, and mobility. J Strength Cond Res. 2014 Aug;28(8):2088-96. doi: 10.1519/JSC.0000000000000258. PMID 25057845
- [Result] Cadore EL, Izquierdo M, Conceicao M, Radaelli R, Pinto RS, Baroni BM, Vaz MA, Alberton CL, Pinto SS, Cunha G, Bottaro M, Kruel LF. Echo intensity is associated with skeletal muscle power and cardiovascular performance in elderly men. Exp Gerontol. 2012 Jun;47(6):473-8. doi: 10.1016/j.exger.2012.04.002. Epub 2012 Apr 14. PMID 22525196
- [Result] Cesari M, Fielding RA, Pahor M, Goodpaster B, Hellerstein M, van Kan GA, Anker SD, Rutkove S, Vrijbloed JW, Isaac M, Rolland Y, M'rini C, Aubertin-Leheudre M, Cedarbaum JM, Zamboni M, Sieber CC, Laurent D, Evans WJ, Roubenoff R, Morley JE, Vellas B; International Working Group on Sarcopenia. Biomarkers of sarcopenia in clinical trials-recommendations from the International Working Group on Sarcopenia. J Cachexia Sarcopenia Muscle. 2012 Sep;3(3):181-90. doi: 10.1007/s13539-012-0078-2. Epub 2012 Aug 3. PMID 22865205
- [Result] Csapo R, Alegre LM. Effects of resistance training with moderate vs heavy loads on muscle mass and strength in the elderly: A meta-analysis. Scand J Med Sci Sports. 2016 Sep;26(9):995-1006. doi: 10.1111/sms.12536. Epub 2015 Aug 24. PMID 26302881
- [Result] Charlson ME, Charlson RE, Peterson JC, Marinopoulos SS, Briggs WM, Hollenberg JP. The Charlson comorbidity index is adapted to predict costs of chronic disease in primary care patients. J Clin Epidemiol. 2008 Dec;61(12):1234-1240. doi: 10.1016/j.jclinepi.2008.01.006. Epub 2008 Jul 10. PMID 18619805
- [Result] Cho KH, Lee HJ, Lee WH. Intra- and inter-rater reliabilities of measurement of ultrasound imaging for muscle thickness and pennation angle of tibialis anterior muscle in stroke patients. Top Stroke Rehabil. 2017 Jul;24(5):368-373. doi: 10.1080/10749357.2017.1285745. Epub 2017 Feb 15. PMID 28198659
- [Result] Chumlea WC, Cesari M, Evans WJ, Ferrucci L, Fielding RA, Pahor M, Studenski S, Vellas B; International Working Group on Sarcopenia Task Force Members. Sarcopenia: designing phase IIB trials. J Nutr Health Aging. 2011 Jun;15(6):450-5. doi: 10.1007/s12603-011-0092-7. PMID 21623466
- [Result] Cooper C, Fielding R, Visser M, van Loon LJ, Rolland Y, Orwoll E, Reid K, Boonen S, Dere W, Epstein S, Mitlak B, Tsouderos Y, Sayer AA, Rizzoli R, Reginster JY, Kanis JA. Tools in the assessment of sarcopenia. Calcif Tissue Int. 2013 Sep;93(3):201-10. doi: 10.1007/s00223-013-9757-z. Epub 2013 Jul 11. PMID 23842964
- [Result] Cruz-Jentoft AJ, Baeyens JP, Bauer JM, Boirie Y, Cederholm T, Landi F, Martin FC, Michel JP, Rolland Y, Schneider SM, Topinkova E, Vandewoude M, Zamboni M; European Working Group on Sarcopenia in Older People. Sarcopenia: European consensus on definition and diagnosis: Report of the European Working Group on Sarcopenia in Older People. Age Ageing. 2010 Jul;39(4):412-23. doi: 10.1093/ageing/afq034. Epub 2010 Apr 13. PMID 20392703
- [Result] D'Hoore W, Sicotte C, Tilquin C. Risk adjustment in outcome assessment: the Charlson comorbidity index. Methods Inf Med. 1993 Nov;32(5):382-7. PMID 8295545
- [Result] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Result] Fukumoto Y, Ikezoe T, Yamada Y, Tsukagoshi R, Nakamura M, Mori N, Kimura M, Ichihashi N. Skeletal muscle quality assessed from echo intensity is associated with muscle strength of middle-aged and elderly persons. Eur J Appl Physiol. 2012 Apr;112(4):1519-25. doi: 10.1007/s00421-011-2099-5. Epub 2011 Aug 17. PMID 21847576
- [Result] Hodges PW, Pengel LH, Herbert RD, Gandevia SC. Measurement of muscle contraction with ultrasound imaging. Muscle Nerve. 2003 Jun;27(6):682-92. doi: 10.1002/mus.10375. PMID 12766979
- [Result] Iannuzzi-Sucich M, Prestwood KM, Kenny AM. Prevalence of sarcopenia and predictors of skeletal muscle mass in healthy, older men and women. J Gerontol A Biol Sci Med Sci. 2002 Dec;57(12):M772-7. doi: 10.1093/gerona/57.12.m772. PMID 12456735
- [Result] Janssen I, Heymsfield SB, Wang ZM, Ross R. Skeletal muscle mass and distribution in 468 men and women aged 18-88 yr. J Appl Physiol (1985). 2000 Jul;89(1):81-8. doi: 10.1152/jappl.2000.89.1.81. PMID 10904038
- [Result] Katula JA, Rejeski WJ, Marsh AP. Enhancing quality of life in older adults: a comparison of muscular strength and power training. Health Qual Life Outcomes. 2008 Jun 13;6:45. doi: 10.1186/1477-7525-6-45. PMID 18554394
- [Result] Kohrt WM, Bloomfield SA, Little KD, Nelson ME, Yingling VR; American College of Sports Medicine. American College of Sports Medicine Position Stand: physical activity and bone health. Med Sci Sports Exerc. 2004 Nov;36(11):1985-96. doi: 10.1249/01.mss.0000142662.21767.58. No abstract available. PMID 15514517
- [Result] Lambert CP, Evans WJ. Effects of aging and resistance exercise on determinants of muscle strength. J Am Aging Assoc. 2002 Apr;25(2):73-8. doi: 10.1007/s11357-002-0005-0. PMID 23604898
- [Result] Massy-Westropp NM, Gill TK, Taylor AW, Bohannon RW, Hill CL. Hand Grip Strength: age and gender stratified normative data in a population-based study. BMC Res Notes. 2011 Apr 14;4:127. doi: 10.1186/1756-0500-4-127. PMID 21492469
- [Result] McKee PA, Castelli WP, McNamara PM, Kannel WB. The natural history of congestive heart failure: the Framingham study. N Engl J Med. 1971 Dec 23;285(26):1441-6. doi: 10.1056/NEJM197112232852601. No abstract available. PMID 5122894
- [Result] Moreira L, Fronza FC, dos Santos RN, Teixeira LR, Kruel LF, Lazaretti-Castro M. High-intensity aquatic exercises (HydrOS) improve physical function and reduce falls among postmenopausal women. Menopause. 2013 Oct;20(10):1012-9. doi: 10.1097/GME.0b013e3182850138. PMID 23531689
- [Result] Narici MV, Flueck M, Koesters A, Gimpl M, Reifberger A, Seynnes OR, Niebauer J, Rittweger J, Mueller E. Skeletal muscle remodeling in response to alpine skiing training in older individuals. Scand J Med Sci Sports. 2011 Aug;21 Suppl 1:23-8. doi: 10.1111/j.1600-0838.2011.01338.x. PMID 21679320
- [Result] Narici MV, Maganaris CN, Reeves ND, Capodaglio P. Effect of aging on human muscle architecture. J Appl Physiol (1985). 2003 Dec;95(6):2229-34. doi: 10.1152/japplphysiol.00433.2003. Epub 2003 Jul 3. PMID 12844499
- [Result] Pijnappels M, Reeves ND, Maganaris CN, van Dieen JH. Tripping without falling; lower limb strength, a limitation for balance recovery and a target for training in the elderly. J Electromyogr Kinesiol. 2008 Apr;18(2):188-96. doi: 10.1016/j.jelekin.2007.06.004. Epub 2007 Aug 29. PMID 17761436
- [Result] Pillen S, Tak RO, Zwarts MJ, Lammens MM, Verrijp KN, Arts IM, van der Laak JA, Hoogerbrugge PM, van Engelen BG, Verrips A. Skeletal muscle ultrasound: correlation between fibrous tissue and echo intensity. Ultrasound Med Biol. 2009 Mar;35(3):443-6. doi: 10.1016/j.ultrasmedbio.2008.09.016. Epub 2008 Dec 10. PMID 19081667
- [Result] Rizzoli R, Reginster JY, Arnal JF, Bautmans I, Beaudart C, Bischoff-Ferrari H, Biver E, Boonen S, Brandi ML, Chines A, Cooper C, Epstein S, Fielding RA, Goodpaster B, Kanis JA, Kaufman JM, Laslop A, Malafarina V, Manas LR, Mitlak BH, Oreffo RO, Petermans J, Reid K, Rolland Y, Sayer AA, Tsouderos Y, Visser M, Bruyere O. Quality of life in sarcopenia and frailty. Calcif Tissue Int. 2013 Aug;93(2):101-20. doi: 10.1007/s00223-013-9758-y. Epub 2013 Jul 5. PMID 23828275
- [Result] Rutherford OM, Jones DA. Measurement of fibre pennation using ultrasound in the human quadriceps in vivo. Eur J Appl Physiol Occup Physiol. 1992;65(5):433-7. doi: 10.1007/BF00243510. PMID 1425649
- [Result] Seguin R, Nelson ME. The benefits of strength training for older adults. Am J Prev Med. 2003 Oct;25(3 Suppl 2):141-9. doi: 10.1016/s0749-3797(03)00177-6. PMID 14552938
- [Result] Simmons V, Hansen PD. Effectiveness of water exercise on postural mobility in the well elderly: an experimental study on balance enhancement. J Gerontol A Biol Sci Med Sci. 1996 Sep;51(5):M233-8. doi: 10.1093/gerona/51a.5.m233. PMID 8808995
- [Result] Sipila S, Suominen H. Ultrasound imaging of the quadriceps muscle in elderly athletes and untrained men. Muscle Nerve. 1991 Jun;14(6):527-33. doi: 10.1002/mus.880140607. PMID 1852160
- [Result] Sipila S, Suominen H. Knee extension strength and walking speed in relation to quadriceps muscle composition and training in elderly women. Clin Physiol. 1994 Jul;14(4):433-42. doi: 10.1111/j.1475-097x.1994.tb00402.x. PMID 7955941
- [Result] Ticinesi A, Meschi T, Narici MV, Lauretani F, Maggio M. Muscle Ultrasound and Sarcopenia in Older Individuals: A Clinical Perspective. J Am Med Dir Assoc. 2017 Apr 1;18(4):290-300. doi: 10.1016/j.jamda.2016.11.013. Epub 2017 Feb 13. PMID 28202349
- [Result] Tosovic D, Muirhead JC, Brown JM, Woodley SJ. Anatomy of the long head of biceps femoris: An ultrasound study. Clin Anat. 2016 Sep;29(6):738-45. doi: 10.1002/ca.22718. Epub 2016 Jun 13. PMID 27012306
- [Result] Watanabe Y, Yamada Y, Fukumoto Y, Ishihara T, Yokoyama K, Yoshida T, Miyake M, Yamagata E, Kimura M. Echo intensity obtained from ultrasonography images reflecting muscle strength in elderly men. Clin Interv Aging. 2013;8:993-8. doi: 10.2147/CIA.S47263. Epub 2013 Jul 25. PMID 23926426